CLINICAL TRIAL: NCT01271998
Title: Pulmonary Disposition of TR-700 Following Once-Daily Oral 200 mg TR-701 Free Acid in Healthy Volunteers
Brief Title: Pulmonary Disposition of TR-700 Following Once-Daily Oral 200 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-027; TR701-119 (Other: TriusRX Unique ID)
Record Dates: First submitted 2010-12-07; First posted 2011-01-07 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Bacterial Infection
Keywords: antibiotic; healthy subjects; pharmacokinetics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteer (Experimental): healthy volunteers
  Interventions: Drug: TR-701 FA

INTERVENTIONS:
Drug: TR-701 FA — 200 mg, oral, once daily for 3 days.

SUMMARY:
The primary purpose of this study is to determine the steady-state plasma pharmacokinetics (PK) and properties of TR-700 into the pulmonary epithelial lining fluid (ELF) and alveolar macrophages (AM) of healthy volunteers.

DETAILED DESCRIPTION:
No applicable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, between 18 and 55 years of age, inclusive
* Females must be nonpregnant, nonlactating, and either postmenopausal or surgically sterile or practicing an effective method of birth control
* Males must be surgically sterile, abstinent, or practicing an effective method of birth control
* BMI between 20 and 34.9 kg/m2, inclusive

Exclusion Criteria:

* Allergy to lidocaine, midazolam, or other anesthetics/sedatives of similar classes
* Physician-diagnosed migraine headaches within 3 years
* Previous enrollment in a TR-701 or TR-701 FA trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2011-01-03 (Actual); Study Completion 2011-01-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters from plasma. | Day 3
  Pharmacokinetic parameters compared with baseline measurements.

CONTACTS AND LOCATIONS:
Overall Officials: David Nicolau, PharmD, Principal Investigator — Center for Anti-Infective Research and Development
Locations (1):
- Trius Investigator Site 001, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Housman ST, Pope JS, Russomanno J, Salerno E, Shore E, Kuti JL, Nicolau DP. Pulmonary disposition of tedizolid following administration of once-daily oral 200-milligram tedizolid phosphate in healthy adult volunteers. Antimicrob Agents Chemother. 2012 May;56(5):2627-34. doi: 10.1128/AAC.05354-11. Epub 2012 Feb 13. PMID 22330925